CLINICAL TRIAL: NCT06893328
Title: PMNTRWS: A Non-interventional Study on Treatment and Therapeutic Efficacy in Chinese Patients With Primary Membranous Nephropathy (PMNTRWS)"
Brief Title: A Real World Study About PMN
Acronym: PMNTRWS
Status: Recruiting | Type: Observational
Sponsor: Wei Chen (Other)
Responsible Party: Sponsor-Investigator, Wei Chen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: CR2023588-1
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Primary Membranous Nephropathy
Keywords: Real-world Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators designed a randomized, controlled, multicenter clinical study to compare the efficacy and safety of rituximab combined with hormones versus rituximab monotherapy in the treatment of primary membranous nephropathy. At the same time, the investigators conducted a real-world study on patients who did not meet the inclusion and exclusion criteria or were unwilling to enter the RCT cohort, to further observe the trial results in a broader population.

DETAILED DESCRIPTION:
Outcomes

* Primary objective Treatment of primary membranous nephropathy with conventional clinical protocols and observation of its effectiveness and safety in a wide population.
* Exploratory purpose

  1. Evaluate the genome-wide changes in kidney and peripheral blood during treatment.
  2. To evaluate the changes in the single-cell transcriptome of the kidney and peripheral blood during treatment.
  3. Evaluate the changes in the RNA transcriptome of the kidney and peripheral blood during treatment.
  4. Evaluate the changes in the renal and peripheral blood proteome during treatment.
  5. Assess the changes in the metabolome during treatment.
  6. Assess changes in the microbiome during treatment.
  7. Predict the effective population of rituximab by baseline renal pathological images.
* Primary outcome The complete response rate at 12 months;
* Secondary outcomes

  1. Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response);
  2. Median remission time;
  3. Proportion of patients without recurrence at 12, 18 and 24 months;
  4. Median non-recurrence time;
  5. Cumulative dose of glucocorticoids;
  6. CD19+ cell count, anti-PLA2R antibody expression level;
  7. Renal function index: eGFR;
  8. Incidence of adverse events;

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as primary membranous nephropathy (PMN) by renal biopsy; 2. Aged over 18 years; 3. An average 24-hour urine protein ≥ 3.5g twice a week after treatment with ACE inhibitors or ARBs for at least 3 months.

-

Exclusion Criteria:

1. With secondary membranous nephropathy (such as hepatitis B and C, systemic lupus erythematosus, drug therapy, malignant tumors and other secondary causes);
2. Active infection, such as active hepatitis B or hepatitis C, tuberculosis (evidence of active tuberculosis infection within 1 year), or human immunodeficiency virus HIV infection (positive for anti-HIV antibodies), etc.
3. A history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or organ transplantation.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as primary membranous nephropathy (PMN) by renal biopsy, with indications for immunosuppressive therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
The complete response rate at 12 months | 12 months
  The complete response rate at 12 months

SECONDARY OUTCOMES:
Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response) | 24 months
  Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response)
Median remission time | 24 months
  Median remission time
Proportion of patients without recurrence at 12, 18 and 24 months | 24 months
  Proportion of patients without recurrence at 12, 18 and 24 months
Median non-recurrence time | 24 months
  Median non-recurrence time
Cumulative dose of glucocorticoids | 24 months
  Cumulative dose of glucocorticoids
CD19+ cell count, anti-PLA2R antibody expression level | 24 months
  CD19+ cell count, anti-PLA2R antibody expression level
Renal function index: eGFR | 24 months
  Renal function index: eGFR
Incidence of adverse events | 24 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Chen, Guangzhou, Guangdong, China